CLINICAL TRIAL: NCT04405739
Title: The Safety of EIDD-2801 and Its Effect on Viral Shedding of SARS-CoV-2
Brief Title: The Safety of Molnupiravir (EIDD-2801) and Its Effect on Viral Shedding of SARS-CoV-2 (END-COVID)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ridgeback Biotherapeutics, LP (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EIDD-2801-2004
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV 2
MeSH Terms: interventions — molnupiravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EIDD-2801 twice daily (BID) for 5 days (Experimental): EIDD-2801 orally twice daily (BID) for 5 days at Dose A, Dose B, Dose C, Dose D, Dose E, Dose F
  Interventions: Drug: EIDD-2801
- placebo (PBO) twice daily (BID) for 5 days (Placebo Comparator): Placebo (PBO) orally twice daily (BID) for 5 days matched for size and appearance to active IP
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EIDD-2801 — Oral capsule of EIDD-2801
  Other Names: molnupiravir; MK-4482
  Arms: EIDD-2801 twice daily (BID) for 5 days
Drug: Placebo — Oral placebo capsule
  Other Names: PBO
  Arms: placebo (PBO) twice daily (BID) for 5 days

SUMMARY:
Designed as a multi-center, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of EIDD-2801 on SARS-CoV-2 Virus Shedding in Newly Hospitalized Adults with polymerase chain reaction (PCR)-Confirmed COVID-19.

DETAILED DESCRIPTION:
Phase 2a randomized, placebo-controlled, double-blinded clinical trial of EIDD-2801 (also known as MK 4482) in adult men and women who have tested positive for severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) infection by polymerase chain reaction (PCR) test within 6 days (144 hours) prior to randomization and are hospitalized with a diagnosis of COVID-19. Rapid enrollment and treatment will be initiated such that the first dose of EIDD-2801 or placebo will be administered as soon as possible and within 7 days of onset of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Has COVID-19 disease, defined by having one or more of the following new symptoms and signs (within 7 days):

   * Fevers OR
   * At least one of the following symptoms: cough, shortness of breath, respiratory rate ≥ 20, radiographic evidence of pneumonia OR
   * Anosmia OR
   * other clinical symptoms or signs of COVID-19 that are not otherwise explained by comorbidities or co-diagnoses
2. PCR+ test for SARS-CoV-2.
3. Has new signs or symptoms of COVID-19 that began ≤7 days of anticipated first dose of study drug.
4. Persons ≥18 years old.
5. at the time of first dose.

5. ≥18 years old.

6. Is willing and able to comply with all study procedures including providing informed consent, collection of virology samples, and any safety tests that are not included as part of standard of care (SOC).

7. Is willing and able to take oral medications, and is anticipated to be able to take the full course of 5 days of study drug.

Pregnancy and Contraception: In nonclinical developmental and reproductive toxicity studies, developmental toxicity including malformation was observed in fetuses from pregnant animals dosed with EIDD-2801 (MK 4482). Therefore, treatment with EIDD-2801 is contraindicated in women who are pregnant or nursing and in the male partners of women who are pregnant. Extreme care must be taken to avoid pregnancy during the study and for 4 days after completion of EIDD 2801 dosing in female participants and for 4 days after completion of EIDD-2801 dosing in female partners of male participants.

8. A female participant is eligible to participate if she is not pregnant or breastfeeding and at least one of the following conditions applies:

* Is not a woman of childbearing potential (WOCBP) OR
* Is a WOCBP and using a contraceptive method that is highly effective (a low user dependency method OR a user-dependent method in combination with a barrier method), or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis), as described in Appendix 2 during the intervention period and for at least 4 days after the last dose of study intervention. The investigator should evaluate the potential for contraceptive method failure (ie, noncompliance, recently initiated) in relationship to the first dose of study intervention.
* A WOCBP must have a negative highly sensitive pregnancy test (serum test is required) within 24 hours before the first dose of study intervention.
* Additional requirements for pregnancy testing during and after study intervention are located in Section 4.4.
* The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Given the elevated risk of venous thrombotic events in patients hospitalized with COVID 19 (Benson et al 2020; Spratt et al 2020), estrogen-containing contraceptives must not be started to fulfill the contraceptive requirement of this study at any time during participant's hospitalization. If contraceptives are interrupted as standard of care management of COVID-19 patients and resumed at a later time point, such as at hospital discharge, then abstinence must be practiced for the defined period of back-up contraception per the contraceptive product labeling. After this period, contraceptive use must adhere to Appendix 2.

  9. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 4 days after the last dose of study intervention:
* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
* Must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause [Appendix 2]) as detailed below:

Agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a WOCBP who is not currently pregnant. Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.

• Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. Is anticipated to require ICU admission for mechanical ventilation within 24 hours of enrollment.
2. Requires more than 6 liters/minute of oxygen to maintain O2 saturation above 95%
3. Is not expected to survive longer than 24 hours.
4. Has a platelet count less than 100,000/µL, hemoglobin less than 9 g/dL, or has a disorder of the hematologic system including anemic disorder or other blood dyscrasia, cancer of the hematologic system, history of bone marrow transplant, or other significant hematologic disease.
5. Women who are pregnant or breastfeeding.
6. Is experiencing DAIDS AE grading scale grade 4 baseline medical conditions or laboratory abnormalities..
7. Has received a vaccine for COVID-19 prior to enrollment, or plans to receive a vaccine for COVID-19 before the end-of-study visit.
8. Has received an experimental antiviral treatment for COVID-19 prior to enrollment.
9. Has received convalescent plasma or other monoclonal antibodies prior to enrollment..
10. Is participating in another clinical study that involves pharmacologic intervention or has participated in another study within 30 days of 5 half-lives of the investigational agent (observational study participation is permitted).
11. In the opinion of the investigator, has end-organ disease as a result of relevant comorbidities: chronic kidney disease (reduced glomerular filtration rate (GFR) <30 mL/min by the Modification of Diet in Renal Disease (MDRD) study equation prior to COVID-19 symptom onset), decompensated chronic liver disease or cirrhosis, decompensated congestive heart failure, active peripheral vascular disease including active diabetic ulcers, chronic pulmonary disease prior to COVID-19 symptom onset requiring bilevel positive airway pressure (BiPAP) or >4 L/min supplemental oxygen at baseline; if using ≤4 L/min supplemental oxygen at baseline, consultation with and approval of the sponsor is required prior to enrollment.
12. Has a diagnosis of cancer that is not in remission. Noninvasive cancers, such as basal and squamous cell carcinoma or history of in situ tumors are allowed at the discretion of the investigator after discussion with the sponsor.
13. Has received an organ transplantation.
14. Has received a bone marrow transplantation.
15. Has been on immunosuppressive medications within one month prior to enrollment.
16. Has any condition that would, in the opinion of the investigator, put the participant at increased risk for participation in a clinical trial.
17. Has known active hepatitis C (HCV RNA positive), active hepatitis B (hepatitis B surface antigen positive), or HIV (ELISA and confirmatory Western blotting). New screening tests not required.
18. Is currently taking nucleos(t)ide analogues for HIV or Hepatitis B, or for their prevention, within 30 days of study enrollment.
19. Is currently taking systemic corticosteroids other than replacement doses, or for treatment of COVID-19.
20. Has a Body Mass Index (BMI) >50 kg/m2.
21. Is anticipated to require surgery within 48 hours after hospital admission.
22. Is anticipated to have a nothing per mouth (NPO) order placed within 48 hours after hospital admission that is expected to last for > 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Balagopal, MD, Principal Investigator — Johns Hopkins University
Locations (11):
- United States (11):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Cook County Hospital, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Ochsner LSU Health Shreveport Academic Medical Center, Shreveport, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - John Hopkins Hospital, Baltimore, Maryland
  - Howard County General Hospital, Columbia, Maryland
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Cox RM, Wolf JD, Plemper RK. Therapeutically administered ribonucleoside analogue MK-4482/EIDD-2801 blocks SARS-CoV-2 transmission in ferrets. Nat Microbiol. 2021 Jan;6(1):11-18. doi: 10.1038/s41564-020-00835-2. Epub 2020 Dec 3. PMID 33273742

RESULTS

PARTICIPANT FLOW:
Groups:
- Molnupiravir 200 mg; Molnupiravir 400 mg; Molnupiravir 800 mg: molnupiravir twice daily (BID) for 5 days
- Placebo: Placebo twice daily (BID) for 5 days
Period: Overall Study
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
Started | 4 | 18 | 25 | 24
Completed | 4 (Molnupiravir 200-mg arm includes 1 participant randomized to molnupiravir 300 mg under protocol version 2) | 13 | 22 | 18
Not Completed | 0 | 5 | 3 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Transferred to rehab | 0 | 0 | 0 | 1
Not completed — Pt. refused IP after 1 dose | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: molnupiravir twice daily (BID) for 5 days
- Total: Total of all reporting groups
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo | Total
Number analyzed (Participants) | 4 | 18 | 25 | 24 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.07) | 52.1 (16.37) | 53.5 (15.42) | 57.1 (14.43) | 54.5 (14.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 11 | 11 | 28
  Male | 4 | 12 | 14 | 13 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 10 | 11 | 8 | 30
  Not Hispanic or Latino | 3 | 8 | 14 | 16 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 1 | 3
  Black or African American | 2 | 2 | 7 | 4 | 15
  White | 1 | 7 | 12 | 14 | 34
  Unknown/Not reported | 0 | 1 | 0 | 1 | 2
  Other | 1 | 7 | 3 | 4 | 15
  More than one race | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 RNA by qPCR in NP Swabs [Mean (Standard Deviation); unit: log 10 copies/mL] — Population: Baseline SARS-CoV-2 values were missing for participants for whom the qPCR test value fell below the lower limit of quantification.
  log 10 copies/mL
    number analyzed (Participants) | 4 | 15 | 23 | 20 | 62
    (all) | 6.45 (1.655) | 4.83 (1.487) | 4.77 (1.442) | 5.07 (1.553) | 5.24 (0.42)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieve Virologic Clearance After Oral Administration of EIDD-2801
Description: Achievement of undetectable (below the limit of detection of the assay) SARS-CoV-2 RNA by day 5 in NP swabs by quantitative Polymerase Chain Reaction (qPCR) in the Efficacy Analysis Set (EAS). The Efficacy Analysis Set consisted of all participants treated with at least on dose of study drug and with at least 1 post baseline assessment of SARS-CoV-2 RNA in NP swabs by qPCR
Time Frame: 28 days
Population: EAS Population
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
Number analyzed (Participants) | 4 | 16 | 25 | 24
Participants | 0 | 4 | 10 | 7

2. Primary Outcome: Number of Participants With Any Serious Adverse Events(SAEs) as Assessed by DAIDS
Description: Incidence of Serious Adverse Events in subjects receiving EIDD-2801 as assessed by DAIDS in the Safety Population, defined as all participants treated with at least one dose of study drug.
Time Frame: 28 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
Number analyzed (Participants) | 4 | 18 | 25 | 24
Participants | 0 | 0 | 1 | 3

3. Primary Outcome: Number of Participants With Any Adverse Events(AEs) as Assessed by DAIDS
Description: Incidence of Adverse Events in subjects receiving EIDD-2801 as assessed by DAIDS
Time Frame: 28 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
Number analyzed (Participants) | 4 | 18 | 25 | 24
Participants | 4 | 11 | 12 | 15

ADVERSE EVENTS:
Time Frame: 28 days
Description: Adverse event is defined as any undesirable sign, symptom or medical condition occurring after starting the study drug (or therapy/intervention) even if the event is not considered to be related to the study. All AEs experienced by participants will be collected and reported from the first dose of EIDD 2801, throughout the study, and will be followed for 28 days unless related to the investigational agent.
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/18 | 1/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/18 | 1/25 | 3/24
Other Adverse Events (participants affected / at risk) | 4/4 | 11/18 | 8/25 | 12/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molnupiravir 200 mg (N=4) | Molnupiravir 400 mg (N=18) | Molnupiravir 800 mg (N=25) | Placebo (N=24)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molnupiravir 200 mg (N=4) | Molnupiravir 400 mg (N=18) | Molnupiravir 800 mg (N=25) | Placebo (N=24)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is requested to obtain written consent from the Sponsor before anything relating to the study can be published.

DOCUMENTS (2):
  • Study Protocol (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT04405739/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT04405739/SAP_001.pdf